CLINICAL TRIAL: NCT01540812
Title: Treatment of Acute Lymphoblastic Leukemia HIGH RISK BCR / ABL NEGATIVE IN ADULTS
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LAL-AR/2011
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Neoadjuvant Therapy; Daunorubicin; Prednisone; Methotrexate; Cytarabine; Hydrocortisone; Idarubicin; fludarabine; Granulocyte Colony-Stimulating Factor; Dexamethasone; pegaspargase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- V + Dauno+ Pred+ Metot+ Cyta+ Hc + Ida + Flud: Vincristine in induction:5 mg/m2 i.v. days 1, 8, 15 and 22 in induction phase Daunorubicin in induction 45 mg/m2 i.v. days 1, 8, 15 and 22 Prednisone in induction: 60 mg/m2/ day, i.v. o p.o., days 1 to 14; 30 mg/m2/day, i.v. o p.o., days 15 to 21; 15 mg/m2/day i.v. o p.o., days 21 to 28 Metotrexato 12 mg days 1 and 22 (intrathecal) Cytarabine (ARA-C): 30 mg days 1 and 22 (intrathecal) Hydrocortisone: 20 mg days 1 and 22 (intrathecal) Idarubicin-induction 2 12 mg/m2, i.v., days 1, 3 and 5 Fludarabine in induction-2: Fludarabine 30 mg/m2, i.v., days, 1 to 5
  Interventions: Drug: Vincristine in induction; Drug: Daunorubicin in induction; Drug: Prednisone in induction; Drug: Metotrexato in induction; Drug: Cytarabine in induction; Drug: Hydrocortisone in induction; Drug: Idarubicin in induction-2; Drug: Fludarabine in induction-2; Drug: Ara-C in induction-2; Drug: G-CSF in induction-2; Drug: Dexamethasone in consolidation-1; Drug: Vincristrine in consolidation-1; Drug: Metotrexato in consolidation-1; Drug: PEG-ASP in consolidation-1; Drug: Dexamethasone in consolidation-2; Drug: ARA-C in consolidation-2; Drug: PEG-ASP in consolidation-2; Drug: Dexamethasone in consolidation-3; Drug: Vincristine in consolidation-3; Drug: Metotrexato in consolidation-3; Drug: PEG-ASP in consolidation-3; Procedure: allogeneic HSCT; Procedure: Allo HSCT with reduced-intensity conditioning

INTERVENTIONS:
Drug: Vincristine in induction
Drug: Daunorubicin in induction
Drug: Prednisone in induction
Drug: Metotrexato in induction
Drug: Cytarabine in induction
Drug: Hydrocortisone in induction
Drug: Idarubicin in induction-2
Drug: Fludarabine in induction-2
Drug: Ara-C in induction-2
Drug: G-CSF in induction-2
Drug: Dexamethasone in consolidation-1
Drug: Vincristrine in consolidation-1
Drug: Metotrexato in consolidation-1
Drug: PEG-ASP in consolidation-1
Drug: Dexamethasone in consolidation-2
Drug: ARA-C in consolidation-2
Drug: PEG-ASP in consolidation-2
Drug: Dexamethasone in consolidation-3
Drug: Vincristine in consolidation-3
Drug: Metotrexato in consolidation-3
Drug: PEG-ASP in consolidation-3
Procedure: allogeneic HSCT
Procedure: Allo HSCT with reduced-intensity conditioning

SUMMARY:
Trial protocol intended the optimization of induction treatment with:

1. Inclusion of PEG-ASP in induction and in the three blocks of consolidation.
2. Reduction of the dose of daunorubicin, and recent studies have shown that the use of high doses of anthracyclines has not brought higher response rates or longer duration
3. Replacing the poor cytological response at day 14 by the level of ER at the end of induction as a criterion to decide the further treatment (consolidation or second induction), so as to have only one criterion (the ER) throughout the study to decision making.

For another hand, reducing non-essential drugs consolidation blocks to try to reduce toxicity during it, and replace the ASP E. coli in induction and consolidation of PEG-ASP to ensure a more sustained asparagine depletion. Also, increasing the dose of methotrexate (3 to 5 g/m2) in patients with ALL-T, since there is recent evidence of a higher response rate with this strategy.

Performing an allo-HSCT early (after one cycle of consolidation) for patients with inadequate level of ER after two cycles of induction or in those patients who required two courses of induction and have obtained proper ER after the second.

Conducting studies of RD centrally by cytofluorometry following Euroflow consensus standards, to avoid bias in making treatment decisions

ELIGIBILITY:
Inclusion Criteria:

* ALL de novo high-risk criteria
* Age 15-55 years (55-60 years patients will be included at the discretion of the medical team that will attend)
* No prior treatment, except Emergency leukapheresis Emergency treatment of hyperleukocytosis with hydroxyurea Urgent cranial irradiation (one dose) for CNS leukostasis Mediastinal irradiation for urgent superior vena cava syndrome
* General condition suitable scale (ECOG 0-2), or> 2 if due to ALL
* Negative pregnancy test for women of childbearing age
* Written informed consent because, although the protocol does not include the use of investigational drugs, biological samples sent there for them

Exclusion Criteria:

* L3 type ALL or mature phenotype B (sIg +) or cytogenetic abnormalities characteristic of mature B-ALL (t (8; 14), t (2, 8), t (8; 22)). For these patients is available BURKIMAB protocol.
* LAL Ph (BCR-ABL) positive. For these patients have the protocol ALL-Ph-08 (if under 55) or LALOPh (if over 55).
* Lymphoid blast crisis of chronic myeloid leukemia
* Biphenotypic acute leukemia or bilinear according to the criteria of EGIL group
* Undifferentiated acute leukemias
* Patients with a history of coronary artery disease, valvular or hypertensive heart disease, contraindicating the use of anthracyclines
* Patients with chronic phase of activity
* Patients with severe chronic respiratory failure
* Kidney failure due to ALL
* Serious neurological disorder not due to the LAL
* History of pancreatitis
* Pregnancy or breastfeeding
* Mental or psychiatric illness preventing informed consent is given for sending samples or properly follow the study
* General condition affected, not attributable to the ALL

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ALL patients
Sampling Method: Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 2 years
  Improve the results of the protocol ALL-AR-03 with modifications in the study methodology of residual disease: centralized, Biomed protocols and the cut-off - <0.01% - internationally accepted and changes in the induction and consolidation treatment, without altering the overall design

SECONDARY OUTCOMES:
Evaluate CR rate with addition of PEG-ASP in the induction phase | 2 years
Standarization of minimal residual disease | 2 years
  Determination of minimal residual disease in a central laboratory trying to homogenice the results
To assess the toxic mortality | 2 years
  To assess whether the reduction of daunorubicin in induction and changes in the consolidation drugs reduce toxic mortality in patients in complete remission
Assess the proportion of non-responders or slow responders | 2 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Ribera JM, Morgades M, Ciudad J, Montesinos P, Esteve J, Genesca E, Barba P, Ribera J, Garcia-Cadenas I, Moreno MJ, Martinez-Carballeira D, Torrent A, Martinez-Sanchez P, Monsalvo S, Gil C, Tormo M, Artola MT, Cervera M, Gonzalez-Campos J, Rodriguez C, Bermudez A, Novo A, Soria B, Coll R, Amigo ML, Lopez-Martinez A, Fernandez-Martin R, Serrano J, Mercadal S, Cladera A, Gimenez-Conca A, Penarrubia MJ, Abella E, Vall-Llovera F, Hernandez-Rivas JM, Garcia-Guinon A, Bergua JM, de Rueda B, Sanchez-Sanchez MJ, Serrano A, Calbacho M, Alonso N, Mendez-Sanchez JA, Garcia-Boyero R, Olivares M, Barrena S, Zamora L, Granada I, Lhermitte L, Feliu E, Orfao A. Chemotherapy or allogeneic transplantation in high-risk Philadelphia chromosome-negative adult lymphoblastic leukemia. Blood. 2021 Apr 8;137(14):1879-1894. doi: 10.1182/blood.2020007311. PMID 33150388